CLINICAL TRIAL: NCT04769661
Title: Role of Cord Blood Cytokines and Perinatal Factors in Prediction of Retinopathy of Prematurity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rewaa Mohammed, Role of cord blood cytokines and perinatal factors in prediction of retinopathy of prematurity, Assiut University
Other Study IDs: RCPR
Record Dates: First submitted 2021-02-22; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cytokines — Doing cord blood cytokines level in preterm infants

SUMMARY:
Cord blood will be taken after birth for evaluation of cytokines level. At age of 4-6 weeks, we will do fundus examination for babies . Retrograde, we will study the perinatal risk factors in subjects found to have retinopathy. Follow up fundus will be done according to results of the first examination. By this study,we will be able later on to predict whom of preterm infants are more prone to develop retinopathy of prematurity.

DETAILED DESCRIPTION:
All patients will be subjected to the following:

1. Clinical evaluation:

   * History taking including name, sex and age at diagnosis of ROP.
   * Detailed obstetric history [maternal age, type of conception (natural, hormonal or in vitro fertilization), type of delivery (vaginal or cesarean section), single or multiple gestation, pregnancy complications (hypertension, diabetes mellitus, placental abruption, premature rupture of membranes, chorioamnionitis), drug history including steroid treatment received prior to delivery].
   * Neonatal data [Gestational age by weeks calculated from the last menstrual period and confirmed by physical examination, birth weight in grams, Apgar scores at 1 and 5 minutes, weight appropriate or small for gestational age, presence of hypoxia during or after delivery, need for oxygen therapy (mode of delivery, duration, oxygen saturation), presence of clinical sepsis, Respiratory distress syndrome, anemia or the need of blood transfusion].
   * Complete physical examination will be done to all babies including cardiac, chest, abdominal and neurological examination.
2. Laboratory assessment:

A- Routine assessment:

1. Complete blood count (CBC) for the mother.
2. CBC for all infants.

B- Immunological assessment: level of Interleukin-6 and 8, and Tumor necrosis factor-α will be assessed:

Umbilical cord blood will be sampled by venipuncture of umbilical vein at birth under complete aseptic conditions for determination of cytokine level. Cord blood samples will be collected on serum separator tube with gel and then are allowed to clot for 30 minutes at room temperature before centrifugation for 15 minutes at 1000xg. Serum will be removed and stored at ≤ -20 ˚c.till assessment by Lab-scan 3D using Luminex assay multiplex kits

3- Fundus examination After training on fundus examination at ophthalmology department, I will do it for babies. Current guidelines by the American Academy of Ophthalmology and Pediatrics, and American Association for Pediatric Ophthalmology and Strabismus recommend that all infants with gestational age ≤32 weeks or birth weight ≤1500g should be screened for retinopathy of prematurity (ROP). Unnecessary examinations may increase the medical costs for ROP screening. First examination will be done at age of 4 to 6 weeks of age, then every 2-3 weeks until their vessels have grown out to the ora serrate and the retina is considered mature. If ROP is diagnosed, examination will be done every 1-2 weeks according to the severity of the disease. The stage of ROP is the highest stage during all fundus examinations done.

ELIGIBILITY:
Inclusion Criteria:

* gestational age less than 32 weeks Birth weight less than 1.5kg

Exclusion Criteria:

* presence of major congenital anomaly Presence of life threatening conditions

Max Age: 1 Hour | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm babies with the previous eligible criteria who were delivered in Women's health hospital and admitted to neonatal intensive care unit of assiut pediatric hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of retinopathy of prematurity | 1 year
  Measure incidence of retinopathy of prematurity in preterm infants
Association of cord blood cytokines and perinatal factors and retinopathy of prematurity | 1 year
  Discover if association exists between cord blood cytokines and perinatal factors and the occurence of retinopathy of prematurity

CONTACTS AND LOCATIONS:
Overall Officials: yasser farouk, lecturer, Study Director — assiut university children hospital

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make individual participant data (IPD) and related data dictionaries available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year
Access Criteria: Through finding the research on clinical trials.gov
URL: http://rewaamohammed2@yahoo.com

REFERENCES:
- [Background] 1. Zin A, Gole GA. Retinopathy of prematurity-incidence today. Clin Perinatol. 2013;40:185-200. PMID: 23719304 DOI: 10.1016/j.clp.2013.02.001 2. Blencowe H, Lawn JE, Vazquez T, Fielder A, Gilbert C. Preterm-associated visual impairment and estimates of retinopathy of prematurity at regional and global levels for 2010. Pediatr Res. 2013;74(Suppl 1):35-49. Pediatr Res. 2013 Dec;74 Suppl 1(Suppl 1):17-34. doi: 10.1038/pr.2013.204.PMID: 24366461 3. Austeng D, Kallen KB, Ewald UW, Jakobsson PG, Holmstrom GE. Incidence of retinopathy of prematurity in infants born before 27 weeks' gestation in Sweden. Arch Ophthalmol. 2009;127:1315-9. PMID: 19822848 DOI: 10.1001/archophthalmol.2009.244 4. Lynch AM, Wagner BD, Hodges JK, et al. The relationship of the subtypes of preterm birth with retinopathy of prematurity. Am J Obstet Gynecol. 2017;217:354. 9. PMID: 28545834 DOI: 10.1016/j.ajog.2017.05.029